CLINICAL TRIAL: NCT00985686
Title: Evaluation of a Spirituality Informed E-mental Health Intervention (LEAP Project) for Major Depressive Disorder in Adolescents and Young Adults - A Randomized Controlled Pilot Trial
Brief Title: E-Mental Health Adolescent Depression Program (LEAP)
Acronym: LEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patricia Steele (Other)
Collaborators: Alberta Centre for Child, Family & Community Research (Other); Alberta Health Services, Calgary (Other); Mount Royal University (Other); SickKids Foundation (Other); University of Calgary (Other)
Responsible Party: Sponsor-Investigator, Patricia Steele, Executive Director, CINIM, Canadian Institute of Natural and Integrative Medicine
Organization: Canadian Institute of Natural and Integrative Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22549; Ethics ID 22549 (Other: Conjoint Health Research Ethics Board)
Record Dates: First submitted 2009-09-24; First posted 2009-09-28 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Depression
Keywords: e-mental health; Adolescent mental health; Spirituality
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Arm (Experimental): Arm where participants began the LEAP Project intervention upon recruitment for an 8 week period.
  Interventions: Other: LEAP Project
- Waitlist Arm (Active Comparator): Arm where participants received the LEAP Project intervention after an 8 week wait period.
  At 8 weeks, the results from the wait-list arm (no intervention) were compared to the results of the study arm (intervention completed).
  Interventions: Other: LEAP Project

INTERVENTIONS:
Other: LEAP Project — In collaboration with experts from Alberta Health Services, the University of Calgary, and Mount Royal University, the Canadian Institute of Natural and Integrative Medicine (CINIM) has created the LEAP Project, a spirituality informed e-mental health intervention, for young people with major depressive disorders (see Appendix for sample materials). It is an online, eight module, multimedia intervention delivered over eight weeks, requiring a weekly commitment of 2-3 hours. The intervention is non-denominational and avoids a focus on any religious traditions. The program aims to treat depression by guiding depressed young people through an exploration of spiritual concepts and principles.

SUMMARY:
The purpose of this project is to explore the potential value and practicality of an innovative depression intervention for young people. More specifically, the objectives of this project are:

1. to pilot the Internet-based Spirituality Program with depressed young people (age 13-24) in Calgary by:

   1. obtaining preliminary estimates on the impact of the program on the primary outcome of depression severity, and secondary outcomes of spiritual well-being and self-concept.
   2. obtaining preliminary estimates on response rates and remission rates to guide sample size estimations for a full size randomized trial.
   3. evaluating if the suggested research methodology is feasible with respect to recruitment rate, patient burden and clinical implementation to guide design of a full size randomized trial.
2. to gather feedback from depressed young people, their families and referral sources in the community (schools, family physicians, mental health outpatient services) on the perceived value of the program and on ways to eventually make it available as a community resource for others dealing with depression.

DETAILED DESCRIPTION:
Depression in adolescents and young adults is a prevalent illness in Canada and presents a high burden for those affected and their families. In Canada, depressive disorders are on the rise and their onset is occurring earlier in life. There is a growing body of evidence suggesting that spiritual wellness may play a role in depression management and recovery. Considering the limitations of available treatments for depression and the significant burden of the disease there is a need for new treatment options that are safe, effective, affordable and acceptable to young people. Our previous research gives strong support to the idea of using a spiritually based intervention for depression. To our knowledge, no research has been conducted on using spirituality as a self-study intervention in the management of depression in young adults. Over the last two years our team has created a spirituality-based intervention program for adolescent depression. The program could present an innovative and low cost treatment option for young patients with major depression.

ELIGIBILITY:
Inclusion Criteria:

* 13-24 years of age
* meet DSM-IV-TR criteria for major depressive disorder (mild-moderate severity) based on the Children's Depression Rating Scale-Revised or the Hamilton Depression Rating Scale
* ability to comply with study intervention, provision of informed assent and/or parental consent

Exclusion Criteria:

In order to avoid confounding through a change in the use of mood altering substances or therapies and through underlying medical conditions, patients will be excluded for any of the following reasons:

* change in use of pharma-therapeutic or herbal treatment for depression in the last three month OR during the first 2 months of trial participation (mild to moderately depressed patients who have not had a change in their treatment in the last three months will be eligible to participate if it is foreseeable that their current treatment will continue unchanged for the first 2 months of trial participation)
* patients currently undergoing a specific psycho-therapeutic treatment that has been shown to be effective for depression (such as Cognitive Behavioral Therapy (CBT) or Interpersonal Therapy (IPT)) or planning to start such therapy in the next two months
* change in the use of medications that have mood altering effects in the last 3 months OR during the first 2 months of trial participation
* history of bipolar disorder, psychotic disorder or psychotic episodes, personality disorder, multiple suicide attempts; history of ADD/ADHD permitted if stabilized (no longer meets DSM-IV-TR criteria for active ADD/ADHD) for at least 2 months; stabilized treated ADD/ADHD permitted if on regular long acting medication and agree to continue
* uncontrolled medical conditions in the last 3 months (assessed by qualified physician)
* high suicide risk
* DSM-IV-TR diagnosis of substance dependence (except nicotine, caffeine) within past 12-months
* history of tx resistance to ≥ 2 antidepressant medications when treated for an adequate period with a therapeutic dose
* recent deaths in the family

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2010-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Toews, MD, FRCPC, Principal Investigator — Canadian Institute of Natural and Integrative Medicine; Badri Rickhi, MB MD FRCPC, Principal Investigator — Canadian Institute of Natural and Integrative Medicine; Jordan Cohen, MD, FRCPC, Principal Investigator — University of Calgary; Dawne Clark, PhD, Principal Investigator — Mount Royal College; John Griffith, BA MDiv, Principal Investigator — Spiritual Directions; Hude Quan, PhD, Principal Investigator — University of Calgary; Janet Chafe, MSW, RSW, Principal Investigator — Alberta Health services; Sabine Moritz, Bsc MSc, Principal Investigator — Alberta Health services; Patti Paccagnan, RN, BN, ACC, Principal Investigator — Canadian Institute of Natural and Integrative Medicine
Locations (1):
- Canadian Institute of Natural and Integrative Medicine (CINIM), Calgary, Alberta, Canada

REFERENCES:
- [Derived] Rickhi B, Kania-Richmond A, Moritz S, Cohen J, Paccagnan P, Dennis C, Liu M, Malhotra S, Steele P, Toews J. Evaluation of a spirituality informed e-mental health tool as an intervention for major depressive disorder in adolescents and young adults - a randomized controlled pilot trial. BMC Complement Altern Med. 2015 Dec 24;15:450. doi: 10.1186/s12906-015-0968-x. PMID 26702639
- See also: Canadian Institute of Natural and Integrative Medicine (CINIM) — http://www.cinim.org
- See also: The LEAP Project — http://www.leapproject.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Arm, Younger Subgroup: Arm where younger participants (13 to 18 years of age) began the LEAP Project intervention upon recruitment for an 8 week period.
  LEAP Project: In collaboration with experts from Alberta Health Services, the University of Calgary, and Mount Royal University, the Canadian Institute of Natural and Integrative Medicine (CINIM) has created the LEAP Project, a spirituality informed e-mental health intervention, for young people with major depressive disorders (see Appendix for sample materials). It is an online, eight module, multimedia intervention delivered over eight weeks, requiring a weekly commitment of 2-3 hours. The intervention is non-denominational and avoids a focus on any religious traditions. The program aims to treat depression by guiding depressed young people through an exploration of spiritual concepts and principles.
- Study Arm, Older Subgroup: Arm where older participants (19 to 24 years of age) began the LEAP Project intervention upon recruitment for an 8 week period.
  LEAP Project: In collaboration with experts from Alberta Health Services, the University of Calgary, and Mount Royal University, the Canadian Institute of Natural and Integrative Medicine (CINIM) has created the LEAP Project, a spirituality informed e-mental health intervention, for young people with major depressive disorders (see Appendix for sample materials). It is an online, eight module, multimedia intervention delivered over eight weeks, requiring a weekly commitment of 2-3 hours. The intervention is non-denominational and avoids a focus on any religious traditions. The program aims to treat depression by guiding depressed young people through an exploration of spiritual concepts and principles.
- Waitlist Arm, Younger Subgroup: Arm where younger participants (13-18 years of age) received the LEAP Project intervention after an 8 week wait period.
  At 8 weeks, the results from the wait-list arm (no intervention) were compared to the results of the study arm (intervention completed).
  LEAP Project: In collaboration with experts from Alberta Health Services, the University of Calgary, and Mount Royal University, the Canadian Institute of Natural and Integrative Medicine (CINIM) has created the LEAP Project, a spirituality informed e-mental health intervention, for young people with major depressive disorders (see Appendix for sample materials). It is an online, eight module, multimedia intervention delivered over eight weeks, requiring a weekly commitment of 2-3 hours. The intervention is non-denominational and avoids a focus on any religious traditions. The program aims to treat depression by guiding depressed young people through an exploration of spiritual concepts and principles.
- Waitlist Arm, Older Subgroup: Arm where older participants (19 to 24 years of age) received the LEAP Project intervention after an 8 week wait period.
  At 8 weeks, the results from the wait-list arm (no intervention) were compared to the results of the study arm (intervention completed).
  LEAP Project: In collaboration with experts from Alberta Health Services, the University of Calgary, and Mount Royal University, the Canadian Institute of Natural and Integrative Medicine (CINIM) has created the LEAP Project, a spirituality informed e-mental health intervention, for young people with major depressive disorders (see Appendix for sample materials). It is an online, eight module, multimedia intervention delivered over eight weeks, requiring a weekly commitment of 2-3 hours. The intervention is non-denominational and avoids a focus on any religious traditions. The program aims to treat depression by guiding depressed young people through an exploration of spiritual concepts and principles.
Period: Overall Study
Arm/Group | Study Arm, Younger Subgroup | Study Arm, Older Subgroup | Waitlist Arm, Younger Subgroup | Waitlist Arm, Older Subgroup
Started | 18 | 16 | 13 | 16
Visit 1: Baseline Data Collection | 18 | 15 | 13 | 16
Visit 2: Data Collection at 8 Weeks | 18 | 15 | 13 | 16
Visit 3: Data Collection at 16 Weeks | 17 | 15 | 13 | 16
Visit 4: Data Collection at 24 Weeks | 17 | 15 | 13 | 14
Completed | 17 | 15 | 13 | 14
Not Completed | 1 | 1 | 0 | 2
Not completed — Lost to Follow-up | 1 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: For study arm, older subgroup - the sample size indicated is 15 instead of 16 as the one participant dropped out after baseline. As no other data was collected for this participant, the decision of the team was to exclude them from the analysis.
Groups:
- Study Arm, Younger Subgroup: Subgroup of participants 13-18 years of age randomized into the study arm.
- Study Arm, Older Subgroup: Subgroup of participants 19-24 years of age randomized into the study arm.
- Waitlist Arm, Younger Subgroup: Subgroup of participants 13-18 years of age randomized into the waitlist arm.
- Waitlist Arm, Older Subgroup: Subgroup of participants 19-24 years of age randomized into the waitlist arm.
- Total: Total of all reporting groups
Arm/Group | Study Arm, Younger Subgroup | Study Arm, Older Subgroup | Waitlist Arm, Younger Subgroup | Waitlist Arm, Older Subgroup | Total
Number analyzed (Participants) | 18 | 15 | 13 | 16 | 62
Age, Continuous [Mean (Full Range); unit: years] | 15.3 [13 to 18] | 21.0 [19 to 24] | 15.2 [13 to 17] | 20.9 [19 to 24] | 18.1 [13 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 8 | 12 | 10 | 44
  Male | 4 | 7 | 1 | 6 | 18
Region of Enrollment [Number; unit: participants]
  Canada | 18 | 15 | 13 | 16 | 62
Use of other treatments during intervention phase [Number; unit: participants]
  Anti-depressants only | 3 | 4 | 2 | 1 | 10
  Counselling only | 4 | 5 | 3 | 4 | 16
  Anti-depressants and Counselling | 0 | 0 | 1 | 1 | 2
  None | 11 | 6 | 7 | 10 | 34
Education [Number; unit: participants]
  High School | 15 | 0 | 13 | 0 | 28
  Post Secondary Institution | 1 | 10 | 0 | 14 | 25
  Not in School | 2 | 5 | 0 | 2 | 9
Religions denomination indicated [Number; unit: participants]
  Yes | 11 | 6 | 5 | 8 | 30
  No | 7 | 9 | 8 | 8 | 32
Work situation [Number; unit: participants]
  Working | 5 | 8 | 3 | 10 | 26
  Not Working | 13 | 7 | 10 | 6 | 36
Living situation [Number; unit: participants]
  With both parents | 7 | 8 | 8 | 10 | 33
  One parent | 8 | 3 | 3 | 3 | 17
  Partner | 0 | 1 | 0 | 0 | 1
  Roommate | 0 | 2 | 0 | 0 | 2
  Alone | 0 | 1 | 0 | 1 | 2
  Other | 3 | 0 | 2 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Children's Depression Rating Scale Revised (CDRS-R)
Description: Measure of depression severity in individuals 13 to 18 years of age. CDRS-R total raw scores includes the sum of 17 items, each item's scoring range is from 1 (no difficulties) to 5 (severe clinically significant difficulties) or 1 (no difficulties) to 7 (severe clinically significant difficulties), with a total possible raw score ranging from 17 to 113. To meet eligibility requirements, participants required a total raw score of 40 to 70.
Time Frame: At 8 week intervals over a 24 week period
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Younger Subgroup (13-18 Years of Age): Subgroup of participants 13-18 years of age. Participants were randomized into the Study and Waitlist Arms.
Arm/Group | Younger Subgroup (13-18 Years of Age)
Number analyzed (Participants) | 31
units on a scale
  Study Arm - Baseline (n=18) | 57.18 (1.87)
  Waitlist Arm - Baseline (n=13) | 61.67 (2.21)
  Study Arm - Week 8 (n=18) | 44.94 (2.86)
  Waitlist Arm - Week 8 (n=13) | 58.93 (3.37)
  Study Arm - Week 16 (n=18) | 36.54 (2.77)
  Waitlist Arm - Week 16 (n=13) | 44.97 (3.26)
  Study Arm - Week 24 (n=17) | 34.37 (3.22)
  Waitlist Arm - Week 24 (n=13) | 42.28 (3.79)

2. Primary Outcome: Hamilton Depression Rating Scale (HAMD)
Description: Measure of depression severity in individuals 19 to 24 years of age. HAMD total scores includes the sum of 17-items, with eight items scored on a range of 0 (absent) to 2 (marked or definite) and nine scored on a range of 0 (absent) to 4 (very severe). The level of depression was based on the following scoring ranges: 7 or under not depressed, 8-13 some depressive symptoms but no depressive disorder, 12-15 mild depression, 16-19 moderate depression, 20-24 moderately severe depression, and 25+ severe depression. To meet eligibility requirements, participants required a total score of 12-24.
Time Frame: At 8 week intervals over a 24 week period
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Older Subgroup (19-24 Years of Age): Subgroup of participants 19-24 years of age. Participants were randomized into the Study and Waitlist Arms.
Arm/Group | Older Subgroup (19-24 Years of Age)
Number analyzed (Participants) | 31
units on a scale
  Study Arm - Baseline (n=15) | 22.14 (0.65)
  Waitlist Arm - Baseline (n=16) | 20.90 (0.65)
  Study Arm - Week 8 (n=15) | 14.07 (1.13)
  Waitlist Arm - Week 8 (n=16) | 17.79 (1.12)
  Study Arm - Week 16 (n=15) | 11.40 (1.39)
  Waitlist Arm - Week 16 (n=16) | 9.91 (1.39)
  Study Arm - Week 24 (n=15) | 8.81 (1.4)
  Waitlist Arm - Week 24 (n=14) | 8.49 (1.40)

3. Secondary Outcome: Piers-Harris Children's Self-Concept Scale - Second Edition (Piers Harris 2)
Description: Measure of self-concept in 13 to 18 year olds. The scale can be completed in 10-15 minutes and includes 60 items covering six subscales: physical appearance and attributes, intellectual and school status, happiness and satisfaction, freedom from anxiety, behavioural adjustment and popularity.
Time Frame: At 8 week intervals over a 24 week period
Reporting Status: Not Posted

4. Secondary Outcome: Six Factor Self-Concept Scale
Description: Measure of self concept in 19 to 24 year olds. The Six-Factor Self-Concept Scale is a multidimensional measure of adult self-concept that was designed to have broad applicability across life settings, roles, and activities. The scale consist of 115 items and assess six factors including likability, morality, task accomplishment, giftedness, power and vulnerability.
Time Frame: At 8 week intervals over a 24 week period
Reporting Status: Not Posted

5. Secondary Outcome: Profile of Mood States (POMS)
Description: Measure of psychological well-being in 19 to 24 year olds. The POMS has the format of an adjective check list and consists of 65 items. It provides a total score of mood disturbance and six factor based subscale scores.
Time Frame: At 8 week intervals over a 24 week period
Reporting Status: Not Posted

6. Secondary Outcome: Spiritual Well-Being Scale (SWBS)
Description: Measure of level spiritual well-being in 13-18 year olds. The self administered 10-item version was used.
Time Frame: At 8 week intervals over a 24 week period
Reporting Status: Not Posted

7. Secondary Outcome: Spiritual Involvement and Belief Scale (SIBS)
Description: Measure of spiritual well-being in 19 to 24 year olds. The instrument is self-administered and contains 26 items in a Likert-type format.
Time Frame: At 8 week intervals over a 24 week period
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Study Arm, Younger Subgroup: Participants 13-18 years of age randomized into the study group
- Study Arm, Older Subgroup: Participants 19-24 years of age randomized into the study group
- Waitlist Arm, Younger Subgroup: Participants 13-18 years of age randomized into the waitlist group
- Waitlist Arm, Older Subgroup: Participants 19-24 years of age randomized into the wait list group
Arm/Group | Study Arm, Younger Subgroup | Study Arm, Older Subgroup | Waitlist Arm, Younger Subgroup | Waitlist Arm, Older Subgroup
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/15 | 0/13 | 0/16
Other Adverse Events (participants affected / at risk) | 0/18 | 0/15 | 0/13 | 0/16

LIMITATIONS AND CAVEATS:
Limitations Inconsistent followup by all study participants Overall generalizability is limited due to a predominantly female sample Self-selection of participants with an open attitude to spirituality No comparison to placebo or active treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No